CLINICAL TRIAL: NCT01943175
Title: Stem Cell-based Approaches to Neuronal Characteristics and Endophenotype of Schizophrenia in Genetic High Risk Subjects
Brief Title: Stem Cell Research on Subjects at Genetic High Risk for Schizophrenia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor
Other Study IDs: H-1207-117-419; A120476 (Other Grant/Funding Number: Korean Health Technology R&D Project)
Record Dates: First submitted 2013-09-04; First posted 2013-09-16 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2013-12

CONDITIONS: Genetic High Risk for Schizophrenia
Keywords: schizophrenia; stem cells; neurons; genetic hish risk for schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 5-10mL of adipose cells in tumescent solution
  5-10mL of venous blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Genetic High Risk
- Healthy Control

SUMMARY:
This study aims at finding endophenotypes of schizophrenia at neuronal level by obtaining stem cells which is derived from adipose cells of subjects with heavy genetic loading for schizophrenia then differentiating them into neuronal cells.

ELIGIBILITY:
Inclusion Criteria:

[Subjects at genetic high risk for schizophrenia]

* Healthy without any Axis I mental disorder
* Is a monozygotic twin of a patient with schizophrenia OR Has at least two family members of schizophrenia in the pedigree, including at least one 1st-degree family member

[Healthy Control]

* Healthy without any Axis I mental disorder
* No family members of schizophrenia in the pedigree to the 3rd degree

Exclusion Criteria:

* Significant neurological or medical illness
* Psychotic symptoms
* Substance abuse
* Suicidal risk
* Blindness or hearing loss
* Taking aspirin, warfarin or hormonal agents
* Pregnancy or lactation
* Susceptibility for keloid formation
* Allergy to lidocaine
* History of significant head trauma or loss of consciousness
* Mental retardation

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Subjects at genetic high risk for schizophrenia
  * Healthy control
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Structural and functional characteristics of neurons differentiated from adipose tissue derived stem cells in subjects with genetic high risk for schizophrenia and healthy controls | three years
  in vitro measurement of the expression of the neuronal markers for differentiated post-mitotic neuron, GABAergic/Glutamatergic neuron.
  The neuronal connectivity, neurites from soma and synaptic protein levels will be assessed. In addition, RNA and proteins expression (e.g. Glutamate/GABA receptors) , physiological function, and in vitro response to antipsychotics will be evaluated.

SECONDARY OUTCOMES:
CAARMS(Comprehensive assessment of at risk mental states) | Baseline
  Clinical rating scale for prodromal symptoms of psychosis.
PANSS(Positive and Negative Syndrome Scale) | Baseline
  Clinical rating scale for the assessment of symptoms of schizophrenia.
Neurocognitive function test battery (composite) | Baseline
  Neurocognitive function battery comprising tests measuring subjects' intelligence, attention, memory, executive function and social cognitive function.
ERP(event-related potential) profile | Baseline
  ERP profile including P50, P30 & MMN(Mismatch Negativity).
Structural/resting functional MRI data | Baseline
  Structural/resting functional MRI data
Proton MR spectroscopy | Baseline
  Molecular neuroimaging data measuring neurochemical composition profile.
PET imaging data | Baseline
  PET imaging data measuring receptor availability of GABA(gamma-aminobutyric acid) and Glutamate.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea